CLINICAL TRIAL: NCT06392347
Title: Optimizing Scan Efficiency of T1-weighted (T1w) Imaging for Vessel Wall Imaging Protocols
Brief Title: Evaluation of Accelerated Sampling Techniques for Vessel Wall Imaging
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 853628
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Vasculopathy
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to compare and evaluate a faster MR image that has been optimized to look at participants blood vessel walls.

DETAILED DESCRIPTION:
The purpose of this study is to compare and evaluate a faster MR image that has been optimized to look at participants blood vessel walls. This faster MR image technique will image participants blood vessel walls in a shorter period of time and will be compared to the routine MR images that is typically used to image participants blood vessel walls.

The purpose of testing these faster images is to compare the image quality with longer conventional images. The goal is to ensure the investigators maintain high image quality over a shorter period of time. These faster images over a shorter period of time have the advantage of fewer motion-related artifacts.

The hypothesis of this research study is that the compressed sensing (fast acquisition technique) based acquisitions will considerably reduce the scan time and will maintain the diagnostic image quality necessary for the assessment of participants blood vessel walls. Thus, the information gained from this study will help us to determine the efficacy of the accelerated protocols for vessel wall imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age and scheduled to undergo clinical vessel wall MR imaging exams as part of their standard of care.

Exclusion Criteria:

1. Any person under the age of 18
2. Presence of artifact-producing intracranial devices (aneurysm clips/coils, ventricular drains, craniectomy mesh, etc.)
3. Any person with contraindications to MRI (medical instability, non-MRI compatible implanted devices, retained metallic foreign bodies, claustrophobia)
4. Large space-occupying lesions (50 mL) or substantial mass effect (herniation, 5mm midline shift) on preceding brain imaging,
5. Imminently life-threatening co-morbid conditions
6. A history of premorbid disabling neurological or psychiatric disease, current substance abuse or remote substance abuse with permanent organic sequelae
7. Pregnancy or lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The staff will be observant of issues related to undue influence as it relates to any vulnerable populations in the event, they are eligible and enrolled in the study (e.g. there will be no impact on grades, employment status, access to medical care or information). If employees, students, etc. meet the eligibility criteria and are enrolled we will do a thorough and sensitive informed consent process in order to protect their rights and minimize any risk of coercion or undue influence.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2027-08 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Optimizing scan efficiency of T1-weighted (T1w) imaging for vessel wall imaging protocols | 24 months
  The primary outcome of the study will be the raters study where qualitative imaging scores will be provided by experienced radiologists using a four-point scale.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No